CLINICAL TRIAL: NCT05066529
Title: Efficacy of Dry Needling Treatment in Myofascial Pain Syndrome-single Blind Randomized Controlled Trial
Brief Title: Efficacy of Dry Needling Treatment in Myofascial Pain Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Merve Damla Korkmaz, Medical Doctor, Kanuni Sultan Suleyman Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KAEK/2021.03.88
Record Dates: First submitted 2021-08-28; First posted 2021-10-04 (Actual); Last update posted 2021-11-05 (Actual); Status verified 2021-10

CONDITIONS: Trigger Point Pain, Myofascial
Keywords: trigger point; dry-needling; ultrasonography; pain intensity; neck disability
MeSH Terms: conditions — Myofascial Pain Syndromes; Pain | interventions — Dry Needling; Exercise

STUDY DESIGN:
Intervention Model Description: Dry needling is a technique in which a fine needle is used to penetrate the skin, subcutaneous tissues and muscles to mechanically disrupt tissue without the use of anesthesia. Treatment is often used to treat myofascial trigger points.
Who Masked: Investigator, Outcomes Assessor
Masking Description: All treatments will be applied by an investigator and a different blinded investigator will evaluate all participants
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- dry-needling group (Experimental): 32 participants in this group Dry-needling treatment will be applied once a week for three weeks. Servical stretching exercises are given to all participants. (20 repetitions in one session and 2 sessions in a day, three days a week.)
  All participants will be evaluated before treatment, after treatment (at 3rd week) and at 3 month follow-ups.
  Interventions: Procedure: dry-needling
- exercise group (Other): 32 participants in this group Servical stretching exercises are given to all participants. (20 repetitions in one session and 2 sessions in a day, three days a week.)
  All participants will be evaluated before treatment, after treatment (at 3rd week) and at 3 month follow-ups.
  Interventions: Procedure: dry-needling

INTERVENTIONS:
Procedure: dry-needling — Dry needling is a technique in which a fine needle is used to penetrate the skin, subcutaneous tissues and muscles to mechanically disrupt tissue without the use of anesthesia. Treatment is often used to treat myofascial trigger points.
  Other Names: exercise

SUMMARY:
The aim of this study is to investigate the short and long-term effects of dry-needling of participants with trigger points in the upper trapezius muscle.

64 participants who diagnosed with myofascial pain syndrome will be included in the study. All participants will have trigger points in the upper trapezius muscles. They are randomised into two groups: dry needling (n=32) and exercise group (n=32). Ultrasonographic evaluation of trigger points (diameter, circumference and area), pain intensity and neck disability will be evaluated as primary outcome. Active cervical range of motion will be evaluated as secondary outcome.

DETAILED DESCRIPTION:
Objective: The aim of this study is to investigate the short and long-term effects of dry-needling of participants with trigger points in the upper trapezius muscle.

Methods: 64 participants who diagnosed with myofascial pain syndrome will be included in the study. All participants will have trigger points in the upper trapezius muscles. They are randomised into two groups: dry needling (n=32) and exercise group (n=32). Ultrasonographic evaluation of trigger points (diameter, circumference and area), pain intensity and neck disability will be evaluated as primary outcome. Active cervical range of motion will be evaluated as secondary outcome.

All treatments will be applied by an investigator and a different blinded investigator will evaluated all participants. Numerical Rating Scale will be used for evaluating pain intensity and Neck Disability Index will be used for evaluating neck disability.

Dry-needling treatment will be applied once a week for three weeks. Servical stretching exercises are given to all participants. (20 repetitions in one session and 2 sessions in a day, three days a week.)

All participants will be evaluated before treatment, after treatment (at 3rd week) and at 3 month follow-ups.

ELIGIBILITY:
Inclusion Criteria:

* trigger points in the upper trapezius muscle
* 18-45 years old
* no treatment in three months for myofascial pain syndrome (MPS)
* accept to participate treatment program

Exclusion Criteria:

* already treated in 3 months for MPS
* below 18 years and above 45 years old
* no acceptance to participate the trial

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-10-30 (Actual)

PRIMARY OUTCOMES:
diameter of trigger point | 3 month follow-ups
  an ultrasonographic evaluation
circumference of trigger point | 3 month follow-ups
  an ultrasonographic evaluation
area of trigger point | 3 month follow-ups
  an ultrasonographic evaluation
Numerical Rating Scale | 3 month follow-ups
  a questionnaire to evaluate pain intensity
Neck Disability index | 3 month follow-ups
  a questionnaire to evaluate neck disability

SECONDARY OUTCOMES:
active servical range of motion | 3 month follow-ups
  active servical range of motion

CONTACTS AND LOCATIONS:
Overall Officials: Merve Damla Korkmaz, Study Director — Kanuni Sultan Suleyman Training and Research Hospital
Locations (1):
- Kanuni Sultan Suleyman Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Gattie E, Cleland JA, Snodgrass S. The Effectiveness of Trigger Point Dry Needling for Musculoskeletal Conditions by Physical Therapists: A Systematic Review and Meta-analysis. J Orthop Sports Phys Ther. 2017 Mar;47(3):133-149. doi: 10.2519/jospt.2017.7096. Epub 2017 Feb 3. PMID 28158962
- [Result] Gerber LH, Shah J, Rosenberger W, Armstrong K, Turo D, Otto P, Heimur J, Thaker N, Sikdar S. Dry Needling Alters Trigger Points in the Upper Trapezius Muscle and Reduces Pain in Subjects With Chronic Myofascial Pain. PM R. 2015 Jul;7(7):711-718. doi: 10.1016/j.pmrj.2015.01.020. Epub 2015 Feb 4. PMID 25661462
- [Result] Gattie ER, Cleland JA, Snodgrass SJ. Dry Needling for Patients With Neck Pain: Protocol of a Randomized Clinical Trial. JMIR Res Protoc. 2017 Nov 22;6(11):e227. doi: 10.2196/resprot.7980. PMID 29167092